CLINICAL TRIAL: NCT06897553
Title: Acceptance and Commitment Therapy- Based Group Therapy for Mental Health in Neurological Disorders
Brief Title: ACT for Mental Health in Neurological Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bielefeld University (Other)
Responsible Party: Principal Investigator, Simon Ladwig, Research Fellow (Post-Doc), Bielefeld University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-2025-01-13
Record Dates: First submitted 2025-03-18; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Neurological Disorders; Mental Health; Executive Function (Cognition); Depression/Anxiety; Stress; Brain Injury; Post-COVID
Keywords: Acceptance and Commitment Therapy (ACT); group therapy; neurological disorders; brain injury; anxiety; stress; depression; executive functioning; abstraction ability; Post-COVID
MeSH Terms: conditions — Nervous System Diseases; Psychological Well-Being; Depression; Anxiety Disorders; Brain Injuries

STUDY DESIGN:
Intervention Model Description: The study design is adaptive based on the recruitment rate. The study starts with only an intervention condition, in a pre/post design. If recruitment allows for, participants will first enter a waiting list condition over eight weeks and then commence the group therapy (intervention condition). Three assessments take place at start of waiting, start of group therapy (pre) and end of group therapy (post).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Waiting List and ACT group therapy (Experimental): Eight weeks of waiting list are followed by eight weeks of ACT group therapy, see study design.
  Interventions: Behavioral: ACT-based group therapy

INTERVENTIONS:
Behavioral: ACT-based group therapy — ACT-based group therapy based on the manual "Living Well with Neurological Conditions" published by Hill et al. (2017; NHS Fundation Trust; available: https://goo.gl/aX6qB5). The manual was translated into German and adapted by shortening sessions, simplifying language and adapting exercises based on clinical experience. The publication of the feasibility study for the adapted manual is currently in preparation. The group therapy includes eight weekly sessions with a duration of 100 minutes each. Three to six individuals participate in a group. The therapy is delivered by at least one licensed psychotherapists. A co-therapist might be included based on individual needs of the group members.

SUMMARY:
The goal of this clinical trial is to examine the efficacy of this manual for mental health in people with mixed neurological disorders, including post-COVID. These conditions are often associated with cognitive impairment, which may hamper the effects of psychoterapy. Executive functioning and especially the ability to abstract thinking may be useful for individuals using Acceptance and Commitment Therapy. Therefore, the main questions research questions are:

* Is this intervention effective in improving mental health?
* Do executive functions predict the extent of social participation and mental health at the end of therapy? Participants will take part in 8 weekly group therapy sessions of 100 minutes each.

DETAILED DESCRIPTION:
Mental health issues, especially depression, anxiety, and stress, are common in people with neurological disorders and post-COVID but often neglected and hence, remain untreated. Acceptance and Commitment Therapy (ACT) is a promising approach to assist people in adapting to their conditions by improving "psychological flexibility".

A previous study translated an adapted group psychotherapy manual for stroke survivors into German and demonstrated its feasibility. This pilot study also gave first indications on the manual's efficacy in reducing symptoms of anxiety, depression, and stress. The aim of this study is to investigate the efficacy of this ACT-based group therapy. People with neurological disorders may have impairments in executive functions, which can affect the psychotherapeutic process. Since ACT often uses metaphors and imagery, executive functions, particularly the ability to abstract, could influence the efficacy of the therapy and are therefore being investigated in this study. The program includes 8 weekly sessions with a session length of 100 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Value above a cut-off of the DASS-21 subscales (depression > 10, anxiety > 6, and stress > 10)
* Sufficient cognition and language ability (clinical rating)
* Sufficient therapy motivation (clinical rating)

Exclusion Criteria:

* Behavioral disorders (e.g., high irritability or apathy in clinical rating)
* Other severe mental disorder (dementia, psychosis, personality disorders, intellectual disability)
* Simultaneous psychotherapy or neuropsychological therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression and Anxiety Stress Scales-21 (Lovibond, 1995) | Before waiting list condition; and pre- and post-intervention (pre and post are presumably 8 weeks apart)
  Measure of psychological burden to investigate efficacy. Scores range from 0 to 63 with higher values indicating higher burden.
Acceptance and Action Questionnaire-Acquired Brain Injury (Sylvester, 2011) | Before waiting list condition; and pre- and post-intervention (pre and post are presumably 8 weeks apart)
  Measure of psychological flexibility to investigate efficacy. Scores range from 0 to 36 with higher values indicating higher inflexibility.
Wechsler Adult Intelligence Scale - Fourth Edition (Similarities subtest; Wechsler, 2008) | pre- and post-intervention (pre and post are presumably 8 weeks apart)
  Measure of individual's ability to recognize and articulate the commonalities between different objects, reflecting their abstraction ability. This will be used to examine the influence of the ability of abstract thinking. Scores range from 0 to 36 with higher values indicating higher ability of abstraction.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (Kroenke, 2001) | Before waiting list condition; and pre- and post-intervention (pre and post are presumably 8 weeks apart)
  Measure of depressive symptoms to investigate efficacy. Scores range from 0 to 27 with higher values indicating more severe depressive symptoms.
Generalized Anxiety Disorder Scale-7 (GAD-7; Spitzer et al., 2007) | Before waiting list condition; and pre- and post-intervention (pre and post are presumably 8 weeks apart)
  Measure of anxiety symptoms to investigate efficacy. Scores range from 0 to 21 with higher scores indicating higher anxiety.
Valuing Questionnaire (Smout, 2014) | Before waiting list condition; and pre- and post-intervention (pre and post are presumably 8 weeks apart)
  Measure of valued living to investigate efficacy. Scores range from 0 to 60 with higher values indicating higher value-congruent living.
Self-as-context scale (Zettle, 2018) | Before waiting list condition; and pre- and post-intervention (pre and post are presumably 8 weeks apart)
  Measure of self as context to investigate efficacy. Scores range from 10 to 70 with higher values indicating a perspective closer to self-as-context.
World Health Organization Disability Assessment Schedule 2.0 (V.S. Üstün, 2010; Plain German) | Before waiting list condition; and pre- and post-intervention (pre and post are presumably 8 weeks apart)
  Measure of functional impairments and disabilities.
Regensburg Word Fluency Test (Aschenbrenner, 2001) | pre- and post-intervention (pre and post are presumably 8 weeks apart)
  Measure of verbal fluency.
Stroop Test in Vienna Test System (Müller & Ziegler, 2001) | pre- and post-intervention (pre and post are presumably 8 weeks apart)
  Measure of cognitive flexibility and inhibition of irrelevant stimuli.

OTHER OUTCOMES:
Group therapy session questionnaire (Zoubek, 2013; Plain German) | GTS-P Session and GTS-T during the intervention (weekly, after each session), GTS-P Total post-intervention
  Measure of treatment acceptance and satisfaction for patients regarding each session (GTS-P Session), for patients regarding the entire therapy (GTS-P Total), and for therapists regarding the each session (GTS-T).
  GTS-P Session scores from 0 to 24 with higher values indicating higher acceptance.
  GTS-P Total scores from 0 to 8 with higher values indicating higher acceptance. GTS-T scores from 0 to 48 with higher values indicating higher acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Werheid, Prof, Study Chair — Bielefeld University
Locations (1):
- Neuropsychologische Hochschulambulanz Bielefeld, Bielefeld, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on public repository like Mendeley Data, while ensuring that no individual may be identified by the data.
Time Frame: IPD will be available latest six months after completion of data collection, presumably January, 1st, 2027. Data will be deleted after ten years.

REFERENCES:
- [Background] Hill G, Hynd N, Price J, Evans S, Moffitt J, Brechin D. Living Well with Neurological Conditions: An eight-week series of group workshops informed by Acceptance and Commitment Therapy (ACT); 2017. Available from: URL: https://goo.gl/aX6qB5.
- [Background] Bowers H, Hill G, Webster A, Bowman AR. Living well with neurological conditions: Clinical outcomes, insights and reflections on three years of Acceptance and Commitment Therapy group intervention. The Neuropsychologist 2021; 1(12):33-42.